CLINICAL TRIAL: NCT02414204
Title: Phosphodiesterase Type 5 Inhibition to Improve Endothelial Function and Vascular Remodeling in Chronic Kidney Disease and End Stage Renal Disease Patients Requiring New Arteriovenous Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Timmy Lee, MD, Principal investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F150220002
Record Dates: First submitted 2015-04-01; First posted 2015-04-10 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Improve Endothelial Function and Decrease Vascular Stenosis
Keywords: Arteriovenous Fistulas (AVFS); Hemodialysis Fistula Maturation (HFM); Flow-Mediated Dilation (FMD); Nitroglycerin-Mediated (NMD); Venous Plethysmography (VP)
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil (Active Comparator): 20 mg twice a day orally
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo twice a day orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil, a phosphodiesterase 5 inhibitor that enhances the effects of nitric oxide (NO), has been shown in experimental and clinical studies in cardiovascular disease to improve endothelial function and decrease vascular stenosis.
  Arms: Sildenafil
Other: Placebo — Placebo will be over encapsulated to identical to drug comparison
  Arms: Placebo

SUMMARY:
Patients with stage IV and V chronic kidney disease and end stage renal disease requiring hemodialysis at University of Alabama at Birmingham (UAB) Dialysis Clinics will be recruited from the UAB Vascular Access Clinic, which has been the site for recruitment of patients requiring new vascular access for the last 10 years.

DETAILED DESCRIPTION:
The main purpose of this research study is to conduct a research study to determine if Sildenafil compared to placebo will improve the vascular health of arteries and veins before arteriovenous fistula creation (shunt) and how quickly your veins and arteries dilate and increase in blood flow after fistula creation. An arteriovenous fistula (shunt) is a connection between the artery and vein in the arm for dialysis use. Another purpose of this study is to determine if Sildenafil reduces the blood and tissue levels of oxidants prior to fistula creation. Oxidants are harmful substances in the body that damage the cells tissues, and organs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years of age male or female
2. Chronic Kidney Disease Stage IV or V patients or End Stage Renal Disease Patient requiring arteriovenous fistula surgery

Exclusion Criteria:

1. Patient currently on nitrate therapy or any nitric oxide donor in any form
2. Patient currently on protease inhibitor or non-nucleoside reverse transcriptase inhibitor
3. Patient with resting systolic blood pressure <90 mm Hg and diastolic blood pressure < 50 mm Hg.
4. Patient life expectancy < nine months.
5. Patient unable or unwilling to meet study requirements.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timmy Lee, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline and 2 Week FMD/VP Measurements Between Sildenafil Group and Placebo Group
Description: For flow mediated dilation studies (FMD), the brachial artery diameter was measured by ultrasound at baseline. An automated floor pressure cuff was inflated on the upper arm to a suprasystolic pressure that was sustained for 5 minutes, and the brachial diameter measurement was repeated 55-65 seconds after releasing the cuff. FMD was calculated as the percentage change in arterial diameter from baseline.
  For venous occlusion plethysmography studies (VP), forearm volume was measured using a strain-gauge plethysmography device during application of an upper arm BP cuff at increasing but subsystolic pressures. Venous capacitance slope was estimated from the volume-pressure relationship and expressed as a percentage increase in volume per millimeters of mercury.
  The change at baseline and 2 weeks in these measurements between the sildenafil and placebo group will be assessed.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: Change in FMD%
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 2 | 2
Change in FMD% | 10.8 (8.0) | 8.6 (2.9)

2. Secondary Outcome: Number of Participants With a Change in Blood Flow Rate
Description: Blood flow of the fistula at 6 weeks is measured with doppler ultrasound and values of the fistula artery and vein are obtained (ml/min). The difference in blood flow rates of the fistula artery and vein between the sildenafil treated group and placebo group will be assessed.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment until 6 weeks following Arteriovenous Fistula (AVF) surgery
Arm/Group | Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
This was a pilot study. Only four participants were recruited during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02414204/Prot_SAP_000.pdf